CLINICAL TRIAL: NCT06023433
Title: Impact of Gingival Crevicular Fluid microRNAs on Orthodontic Tooth Movement: a Split Mouth Study
Brief Title: Impact of Gingival Crevicular Fluid microRNAs on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal Investigator, University of Catania
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 121-26
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Orthodontic Tooth Movement

STUDY DESIGN:
Intervention Model Description: The main objective of the study is to evaluate the impact of orthodontic tooth movement on gingival crevicular fluid miRNAs related to inflammation and osteoclastogenesis.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canines to be distalized (Active Comparator): The canines need distalization after orthodontic upper first premolar asymmetrical extractions.
  Interventions: Device: Elastomeric powerchain
- Controlateral canines (No Intervention): The controlateral canines don't need distalization since the adjacent first premolars are not extracted.

INTERVENTIONS:
Device: Elastomeric powerchain — Canine distalization by engaging the elastomeric power chains onto the canine brackets.
  Arms: Canines to be distalized

SUMMARY:
A split-mouth study is conducted in order to evaluate the impact of orthodontic movement on the expression of gingival crevicular fluid miRNAs related to inflammation and osteoclastogenesis during canine distalization following asymmetrical extraction treatment of upper first premolars.

Samples of gingival crevicular fluid on the mesial and distal side of the canines to be examined will be performed during the baseline and during various follow-ups.

DETAILED DESCRIPTION:
A split-mouth study is conducted in order to evaluate the impact of orthodontic movement on the expression of gingival crevicular fluid miRNAs related to inflammation and osteoclastogenesis during canine distalization following asymmetrical extraction treatment of upper first premolars.

Orthodontic tooth movement induces bone remodeling by various signaling pathways. The variations in miRNAs expression and their impact in inflammation and osteoclastogenesis during the various stages of orthodontic tooth movements is not fully understood.

58 patients requiring asymmetrical upper first premolar extraction for orthodontic purposes have been enrolled for this split-mouth study: the canines to be distalized on the extractive site are considered as the test group, the controlateral canines (on the side without first premolar extraction) areconsidered as normal controls.

ELIGIBILITY:
Inclusion Criteria:

* patients with excellent oral hygiene throughout the study period,
* patients requiring asymmetrical maxillary first premolar extraction so monolateral canine retraction will be performed as a part of the treatment,
* patients available to come back at the clinic at the times of sample collection.

Exclusion Criteria:

* poor oral hygiene and/or bleeding on probing,
* use medications, steroids or other anti-inflammatory medications,
* systemic health problems or smoking.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
miRNAs expression | 6 weeks
  miRNAs expression in the gingival crevicular fluid by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Pubmed

REFERENCES:
- [Derived] Polizzi A, Alibrandi A, Lo Giudice A, Distefano A, Orlando L, Analazi AM, Pizzo G, Volti GL, Isola G. Impact of periodontal microRNAs associated with alveolar bone remodeling during orthodontic tooth movement: a randomized clinical trial. J Transl Med. 2024 Dec 30;22(1):1155. doi: 10.1186/s12967-024-05933-x. PMID 39736760